CLINICAL TRIAL: NCT03193944
Title: Vitamin D Supplementation on Metabolic Syndrome Indicators Among Food Insecure, Vitamin D Deficient Older Adults in Karaj City, Alborz Province, Iran;
Brief Title: Vitamin D Supplementation on Metabolic Syndrome Indicators Among Older Adults, Alborz Province, Iran
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alborz Medical University (Other Government)
Collaborators: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Maryam Zarei, Principal investigator, Alborz Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Abzums.Rec.1395.114
Record Dates: First submitted 2017-06-13; First posted 2017-06-21 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Vitamin D Deficiency; Diabetes Mellitus; Hypertension; Lipid Metabolism Disorders; Obesity, Abdominal
MeSH Terms: conditions — Vitamin D Deficiency; Diabetes Mellitus; Hypertension; Lipid Metabolism Disorders; Obesity, Abdominal | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: A detailed explanation on research design, location and population, sampling technique, sample size, instrument, data collection, data analysis and potential limitations of the study are outlined in the following sections. This study aims to find relationships between food insecurity, vitamin D intakes and its impact on metabolic syndrome among older adults in a city in Alborz province in Iran, known as Karaj. This study has 2 parts; the first part is to determine the prevalence of food insecurity and vitamin D deficiency among older adults in Karaj city. The second part is an intervention study examining effects of vitamin D supplementation on metabolic syndrome (diabetes, obesity, hypertension, and dyslipidaemia) among older adults who has at least have risk factors of metabolic syndrome, food insecure and vitamin D deficient. The intervention group will receive vitamin D supplementation 50000 IU for 8 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Intervention group will receive 50,000 U vitamin D3 per week (equivalent to 1,250 μg) for 8 weeks
  Interventions: Drug: D-vitin, soft gelatin capsule (vitamin D3,50000 IU)
- control group (Placebo Comparator): Control group will receive vitamin D as a placebo. placebo will be identical in appearance taste and odourless.
  Interventions: Drug: Placebo vitamin D3

INTERVENTIONS:
Drug: D-vitin, soft gelatin capsule (vitamin D3,50000 IU) — Intervention group: The respondents in intervention group will receive 50000 vitamin D for 8 weeks. Plus, brochures and pamphlets related to nutrition and health.
  Other Names: cholecalciferol,
  Arms: Intervention group
Drug: Placebo vitamin D3 — vitamin D as a placebo
  Arms: control group

SUMMARY:
General objective: To assess the effect of vitamin D supplementation on metabolic syndrome among food insecure and vitamin D deficient older adults in Karaj city, Alborz province in Iran. A two-arm randomised controlled trial (RCT) will be conducted by recruiting participants. Inclusion Criteria: Food insecure, metabolic syndrome; Vitamin D deficiency Exclusion Criteria: those who are already taking any type of vitamin D supplements, Individuals with a history of allergy, Those subjects with serious medical condition such as cancer, heart attack, stroke, and etc., Intervention group: The intervention will start from 10 of May 2017 to 11 of July 2017 for 2 months. The intervention group will receive 50,000 U vitamin D3 per week (equivalent to 1,250 μg) for 8 weeks plus pamphlets and brochures about nutrition and health at the beginning of the study. Control group: The respondents in control group will receive placebo plus brochures and pamphlets related to nutrition and health at the beginning of the study. The data collection process will identify the older adults for both groups; intervention and control. Consent will be obtained from those who are eligible. Anthropometric measurement (height, weight, body mass index, and waist circumference), blood pressure measurement, blood taking and three-day food record will be obtained during baseline from all study respondents in the intervention and control groups. Primary Output: Achieving 25 (OH) D upper than insufficient serum 25(OH) D level >30 ng/l. Secondary Output: Reduction anthropometry (body mass index (BMI) and waist circumference (WC), Improved Biomarkers indicators (lipid profile, fasting blood fast), improved blood pressure before and after intervention.

DETAILED DESCRIPTION:
This study aims to find relationships between food insecurity, vitamin D intakes and its impact on metabolic syndrome among older adults in a city in Alborz province in Iran, known as Karaj. This study has 2 parts; the first part is to determine the prevalence of food insecurity and vitamin D deficiency among older adults in Karaj city. The second part is an intervention study examining effects of vitamin D supplementation on metabolic syndrome (diabetes, obesity, hypertension, and dyslipidaemia) among older adults who have at least have risk factors of metabolic syndrome, food insecure and vitamin D deficient. The first part; the data collection process will be performed in a few stages. The first stage will be to initiate contacting with the health centres in Karaj city to identify the older adults. Appointments will be set after screening the study subjects who will be eligible. Consent will be obtained from those who were eligible. The preliminary information on demographic data, socioeconomics, food insecurity, dietary intake and sunlight exposure will be collected by using a set of questionnaires. The blood sample for measuring serum 25 (OH) D will be taken the same day as questionnaires were filled.

The second stage: The data collection process will be performed in few stages. The first stage will include of contact with health centres in Karaj city to identify the older adults for both groups; intervention and control. Consent will be obtained from those who will eligible. Anthropometric measurement (height, weight, body mass index, and waist circumference), blood pressure measurement, blood taking and three-day food record will be obtained during baseline from all study respondents in the intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Food insecure,
* Have fit criteria of metabolic syndrome; (WC>90 cm), obesity (BMI≥30 kg/m2), diabetes (FBS>100 mg/dl), high blood pressure (systolic >135 mmHg and diastolic >85 mmHg) and dyslipidaemia (LDL≥ 240 mg/dl, HDL<40 mg/dl, TC≥ 160 mg/dl; TG≥ 200 mg/dl),
* Vitamin D deficient; serum 25(OH) D level <30 ng/ml,
* No use of vitamin D supplementation before 60 days,

Exclusion Criteria:

* An inability or unwillingness to participate,
* Those who are already taking any type of vitamin D supplements,
* Individuals with a history of allergy,
* Those subjects with serious medical condition such as cancer, heart attack, stroke, and etc.,
* Illness that required corticosteroids or insulin,
* Drugs are known to influence vitamin D level; steroids, anti-acids, oestrogen,
* People with conditions that contradict vitamin D supplementation, for example, a history of hypercalcaemia, hepatic disease or renal stones, sarcoidosis, or malignancy,

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Aged from 60 to 80 years old,
Enrollment: 120 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2017-05-10 (Actual); Study Completion 2017-07-10 (Actual)

PRIMARY OUTCOMES:
Achieving 25 (OH) D upper than insufficient serum 25(OH) D level >30 ng/l. | by 2 months
  According to the guidline, vitamin D deficiency will improve by taking vitamin D3 by 2 months.

SECONDARY OUTCOMES:
Reduction anthropometry (BMI and WC), | by 2 months
  Reduction of BMI, WC after 2 months intervention by vitamin D3
Improved Biomarker indicators (lipid profile) | by 2 months
  Reduction of lipid profiles are important for this research after vitamin D3 intervention.
Improved Biomarker indicator FBS | by 2 months
  Reduction of FBS by 2 months intervention via taking vitamin D
Improved blood pressure | by 2 months
  Reduction of blood pressure after taking vitamin D for 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Zarei, Principal Investigator — World Health Organization
Locations (1):
- Maryam Zarei, Karaj, Alborz Province, Iran

IPD SHARING:
Plan to Share IPD: Yes